CLINICAL TRIAL: NCT04515654
Title: Supporting Trans Identities and Occupational Justice Through Narrative Informed Theatre: A Mixed-methods Pilot Study
Brief Title: Supporting Trans Identities and Occupational Justice Through Narrative Informed Theatre: Supporting Trans Identities and Occupational Justice Through Narrative Informed Theatre
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Sally Wasmuth, Asistant Professor OT, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1906677292
Record Dates: First submitted 2020-05-20; First posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Transgenderism; Stigma, Social
Keywords: gender; drama; disability studies; qualitative; stigma; affirmative care; minority health
MeSH Terms: conditions — Transsexualism; Social Stigma; Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Audience participants (Experimental): Community members viewed the performance (intervention) and completed pre/post stigma questionnaire
  Interventions: Other: IDEAS (Identity Evolution and Sharing) Performance

INTERVENTIONS:
Other: IDEAS (Identity Evolution and Sharing) Performance — 60 minute webinar depicting first-hand stories of transgender and gender non-conforming individuals followed by expert panel/talk-back
  Other Names: Performance

SUMMARY:
Importance: Societal stigma gravely impedes occupational justice for trans individuals, producing vast health disparities for this population.

Objective: Test feasibility and impact of an intervention to reduce stigma and improve trans wellbeing Design: Convergent parallel mixed methods Setting: Community/Webinar Participants: 42 audience members and 6 trans interviewees Intervention: Virtual, narrative-informed play reading and moderated discussion about gender diversity and affirmative care Outcomes and Measures: The valid and reliable Acceptance and Action Questionnaire - Stigma (AAQ-S) assesses stigma beliefs; An open-ended qualitative question assesses trans interviewees' experiences

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Acceptance and Action Questionnaire-stigma | 1 week
  The Acceptance and Action Questionnaire - Stigma (AAQ-S) survey

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Purdue University Indianapolis, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No